CLINICAL TRIAL: NCT04622748
Title: An Investigation of Neurocognitive Functions and the Influencing Factors in Recovered Patients With COVID-19
Brief Title: Neurocognitive Functions of Recovered COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute on Drug Dependence, China (Other)
Collaborators: Peking University Sixth Hospital (Other); Wuhan Wuchang Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: NIDD-2020-Neurocognition
Record Dates: First submitted 2020-09-06; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-09

CONDITIONS: Cognition; Covid-19
MeSH Terms: conditions — COVID-19 | interventions — Psychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19: Recovered COVID-19 patients in Wuhan
  Interventions: Behavioral: Trier Social Stress Test
- Healthy Control: Uninfected people in Wuhan
  Interventions: Behavioral: Trier Social Stress Test

INTERVENTIONS:
Behavioral: Trier Social Stress Test — 8-min oral calculation and 5-min speech

SUMMARY:
This study is carried on in Wuchang Hospital in Wuhan, China. The investigators plan to recruit 80 patients with COVID-19 and 80 matched healthy control. Using the design of case-control study, the study aims to assess the neurocognitive functions such as executive function and attentional bias in recovered patients with COVID-19 under normal and stress conditions, and to analyze the influencing factors of neurocognitive functions, such as mental health conditions, inflammation indicators and cardiopulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* Recovered COVID-19 patients or uninfected residents in Wuhan, with an education level above elementary school and are able to complete cognitive tasks;
* Willing to participate in this study and sign informed consent.

Exclusion Criteria:

* Subjects with body temperature> 38°C;
* Subjects who are in menstruation and pregnancy;
* Subjects suffering from cardiopulmonary diseases before the new coronary pneumonia epidemic (such as heart disease, pulmonary hypertension, congestive heart failure, etc.);
* Subjects with severe disturbances in consciousness, cognitive dysfunction, mental disorders, visual and hearing disorders, bone and joint diseases, etc.;
* Subjects with abnormal immune system and severe organ dysfunction (heart, liver, kidney, etc.);
* Subjects who are unwilling to participate in this study and cannot complete all surveys and cognitive function tests.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recovered COVID-19 patients and uninfected residents in Wuhan
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-12-10 (Estimated); Study Completion 2020-12-10 (Estimated)

PRIMARY OUTCOMES:
working memory | 10 minutes
  assessed by the n-back task, including 0-back, 1-back and 2-back
Cognitive flexibility | 3 minutes
  assessed by the trail-making task
Inhibitory control | 10 minutes
  assessed by the stroop task

SECONDARY OUTCOMES:
Attention Bias | 15 minutes
  assessed by the dot-probe task
Serum TNFalpha | 1 day
  Concentration of serum TNFalpha in ng/ml will be assessed by ELISA
Serum IL-6 | 1 day
  Concentration of serum IL-6 in ng/ml will be assessed by ELISA.
CRP | 1 day
  hypersensitive C-reactive protein(hs-CRP) in mg/L will be assessed by Turbidimetric inhibition immuno assay.
Depression | 3-5 minutes
  assessed by Self-Rating Depression Scale, which is consist of 20 items scoring 1 to 4.
Anxiety | 3-5 minutes
  assessed by Self-Rating Anxiety Scale, which is consist of 20 items scoring 1 to 4.
PTSD | 3-5 minutes
  assessed by PTSD Checklist for DSM-5 (PCL-5)
Sleep | 3-5 minutes
  assessed by Pittsburgh sleep quality index (PSQI)
General cognition | 8-10 minutes
  assessed by Montreal - Cognitive Assessment (MoCA)
Cardiopulmonary function 1 | 15 minutes
  maximal inspiration pressure（MIP), maximal expiration pressure（MEP）
Cardiopulmonary function 2 | 10 minutes
  Assessed by the 6-minutes' walk test

OTHER OUTCOMES:
Stress response indicator 1 | Saliva samples will be colleted before stress, 0 minutes and 10 minutes after stress.
  concentration of saliva cortisol stress, assessed by ELISA
Stress response indicator 2 | Assessed before and 0 minute after stress
  Hear rates
Stress response indicator 3 | Assessed before and 0 minute after stress
  Blood pressure before stress and after stress

CONTACTS AND LOCATIONS:
Overall Officials: Lin Lu, Dr., Study Director — National Institute on Drug Dependence, Peking University
Locations (1):
- Wuhan Wuchang Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No